CLINICAL TRIAL: NCT02394379
Title: A Prospective, Post Approval Study to Evaluate the Trulign™ Toric Posterior Chamber Intraocular Lens (IOL)
Brief Title: Post Approval Study to Evaluate the Trulign™ Toric Posterior Chamber IOL
Status: Completed | Type: Observational
Sponsor: Bausch & Lomb Incorporated (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 858
Record Dates: First submitted 2015-03-09; First posted 2015-03-20 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trulign™ Toric IOL: Trulign™ Toric Posterior Chamber IOL is a modified plate haptic lens
  Interventions: Device: Trulign™ Toric IOL

INTERVENTIONS:
Device: Trulign™ Toric IOL — Trulign™ Toric Posterior Chamber IOL is a modified plate haptic lens

SUMMARY:
To evaluate the incidence of IOL vaulting (ie, position change) of the Trulign™ Toric IOL following cataract surgery.

DETAILED DESCRIPTION:
The objective of this post approval safety study is to evaluate the incidence of IOL vaulting (ie, position change) of the Trulign™ Toric IOL following cataract surgery at up to three years post implantation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able and willing to comply with the follow-up schedule
* Subjects must have a clinically documented diagnosis of age-related cataract that is considered amenable to treatment with standard phacoemulsification/extracapsular cataract extraction
* Subjects must require a lens power from 4 to 33 D
* Subjects must have a Best Corrected Visual Acuity (BCVA) equal to or worse than 20/40, with or without a glare source

Exclusion Criteria:

* Subjects with any anterior segment pathology in the study eye likely to increase the risk of complications from phacoemulsification cataract surgery
* Subjects with associated ocular conditions which could affect the stability of the IOL
* Subjects with clinically significant irregular corneal astigmatism in the study eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be chosen from 30-50 clinical sites in the US. All subjects who meet Eligibility Criteria (below) will be consecutively offered enrollment until the site meets the maximum number of enrollees.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-03-19 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically significant IOL vaulting | Up to 3 years
  IOL vaulting is position change such as clinically significant anterior vaulting, clinically significant tilt, and secondary surgical intervention related to such vaulting. The proportion of study eyes experiencing vaulting will be estimated by Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals NA / Bausch & Lomb
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States